CLINICAL TRIAL: NCT00615693
Title: A Multicenter, Single Sequence, Open-label Study to Assess the Tolerability, Safety, and Efficacy of 2 Weeks Oral AEB071 300 mg Twice Daily, Followed by 6 Weeks AEB071 200 mg Twice Daily in the Treatment of Patients With Macular Edema Associated With Non-infectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis
Brief Title: Safety, Tolerability, and Efficacy of AEB071 in the Treatment of Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB071A2211
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2017-02

CONDITIONS: Uveitis; Posterior Uveitis; Panuveitis
Keywords: Uveitis; Macular Edema
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Panuveitis; Macular Edema | interventions — sotrastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of AEB071 as a therapy for uveitis. Vision improvement and reduction in the swelling of retina will be measured for the assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with non-infectious intermediate or posterior uveitis or panuveitis in at least one eye, age 18 to 70 years of age inclusive, who are otherwise in good health
* Macular edema with average central retinal thickness ≥ 250 µm
* A vitreous haze score ≥ 1, but ≤ 3 (based on the National Eye Institute grading system)
* Best Corrected Visual Acuity no worse than 20/400 and no better than 20/40
* Daily prednisone dose < 1 mg/kg

Exclusion Criteria:

* Patients with choroidal neovascularization.
* Patients with the following forms of uveitis:

  1. Serpiginous choroidopathy
  2. Acute multifocal placoid pigment epitheliopathy
  3. White dot retino-choroidopathies (e.g., multiple evanescent white dot syndrome (MEWDS) or multifocal choroiditis)
* Macular edema associated with other ocular disease (e.g., diabetic retinopathy)
* Patients who had a prior vitrectomy
* Any eye condition that may affect the evaluation of visual acuity and retinal thickness
* Concurrent use of certain immunosuppressive agents (specific washout periods for different agents are defined in the protocol)
* Use of systemic medications known to be toxic to the lens, retina, or optic nerve (e.g. deferoxamine, chloroquine, and ethambutol) currently or in the past 6 months
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AEB071 | Baseline/Day 1 to Week 8 (Day 56) (end of study)

SECONDARY OUTCOMES:
Change in the degree of inflammation in the study eye | Baseline/Day 1, Week 8 (Day 56)/end of study
Change in the visual acuity of the study eye | Baseline/Day 1, Week 8 (Day 56)/end of study
Change in macular edema in the study eye | Baseline/Day 1, Week 8 (Day 56)/end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (13):
- United States (13):
  - University of Southern California Doheny Eye Institute, Los Angeles, California
  - University of California, San Francisco, California
  - Colorado Retina Associates, Denver, Colorado
  - University of Miami Miller School of Medicine; Anne Bates Leach Eye Hosptial;Bascom Palmer Eye Institute, Miami, Florida
  - University of South Florida, Eye Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - John Hopkins Hospital/Wilmer Eye Institute, Baltimore, Maryland
  - MERSI, Cambridge, Massachusetts
  - Mayo Clinic Department of Opthalmology, Rochester, Minnesota
  - Cornea and Laser Eye Institute, Teaneck, New Jersey
  - New York Eye and Ear Infirmary, Clinical Research Department, New York, New York
  - Retina Research Centre, Austin, Texas
  - Vitreoretinal Consultants, Houston, Texas

REFERENCES:
- See also: Results for CAEB071A2211 from the Novartis Clinical Trials website. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3540